CLINICAL TRIAL: NCT00451776
Title: Post Operative Hemodynamic Function After Anesthetic Induction With Etomidate for Cardiac Surgery With ECC. A Prospective, Monocentric, Randomised Double Blind Study
Brief Title: Post Operative Hemodynamic Function After Anesthetic Induction With Etomidate for Cardiac Surgery With ECC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Dr Jérôme MOREL, Centre Hospitalier Universitaire de Saint Etienne
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0608119; 2006-007017-21
Record Dates: First submitted 2007-03-22; First posted 2007-03-23 (Estimated); Last update posted 2008-10-31 (Estimated); Status verified 2008-10

CONDITIONS: Cardiac Surgery
Keywords: cardiac surgery; adrenal insufficiency; etomidate; propofol
MeSH Terms: conditions — Adrenal Insufficiency | interventions — Etomidate; Propofol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): patients who received etomidate
  Interventions: Drug: etomidate
- 2 (Active Comparator): patients who received propofol
  Interventions: Drug: propofol

INTERVENTIONS:
Drug: etomidate — patients who received etomidate
  Arms: 1
Drug: propofol — patients who received propofol
  Arms: 2

SUMMARY:
Because of its hemodynamic safety, etomidate is widely used for anaesthesia induction of cardiac surgery. It can also cause adrenal insufficiency during the following 48 hours ( 11 betahydroxylase inhibition ). So it could increase hemodynamic dysfunction caused by the SIRS following cardiopulmonary bypass.

A previous observational study found more adrenal insufficiency and need for vasopressive support therapy in the etomidate group versus another propofol induced group.

The aim of our work is to compare hemodynamic dysfunction following induction with etomidate for cardiac surgery with ECC. The control group would be induced by Propofol. 94 patients would be included.

DETAILED DESCRIPTION:
Information will be given at the anaesthetic consultation, few weeks before planed cardiac surgery. Eligibility and exclusion criteria will be checked. Patient will receive an informative written consent notice and all questions will be answered. A standard pre-operative blood collection will be sampled.

In order to minimize the potential confusing effect of daily cortisol variation, only surgical procedure performed early morning will be considered. The day before surgery definitive inclusion will be decided as the order of procedure is not known before. Only patients operated in the morning will be included because of cortisol daily variations. At this time, consent and information notice will be signed and checked in the medical record.

On the morning of surgery, during venous catheter insertion an additional blood sample will be collected to asses basal cortisolemia.

Randomisation will be carried out centrally after patient operative theatre admission, by phone call from ICU to randomisation office. Hypnotic drug will be prepared in the ICU department next to the operative room and blindly administered to patient ( same volume per weight ). All other anesthetic procedures will be standardised : opioid drugs, vasopressive support, antifibrinolytics and hemodynamic monitoring.

After surgery patients are admitted to surgical ICU. They will undergo standard post operative exams plus two corticotrophin tests and a dosage of SIRS markers ( IL6 and TNF alpha ). These results will only be known at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* age superior to 18 years
* patient which had to be operated for aorto-coronary pass and/or valvular replacement

Exclusion Criteria:

* patient with aortics shrinking
* women pregnant or nursing
* contra-indication to etomidate or diprivan or synacthene
* patient with insufficiency kidney
* patient with infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2007-06; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Time to discharge to vasoactive supportive therapy in the first 48 post operative hours . | 48 hours

SECONDARY OUTCOMES:
Hemodynamic supportive drugs ( I .e : dodutamine and noradrenaline ) doses at different time . | several times
Systematic inflammatory response intensity | 6 hours
Hemodynamic supportive drugs consumption in patients with SIRS sub group | 24 hours
Myocardial infarction incidence in the first 48 postoperative hours . | 48 hours
In hospital mortality | day of hospital coming out

CONTACTS AND LOCATIONS:
Overall Officials: Jérome MOREL, MD, Principal Investigator — Centre Hospitalier Universitaire de Saint Etienne
Locations (1):
- University hospital, Saint-Etienne, France